CLINICAL TRIAL: NCT05330429
Title: A Phase 2, Randomized, Open-Label Study Evaluating the Safety and Efficacy of Magrolimab in Combination With Bevacizumab and FOLFIRI Versus Bevacizumab and FOLFIRI in Previously Treated Advanced Inoperable Metastatic Colorectal Cancer (mCRC)
Brief Title: Study of Magrolimab Given Together With FOLFIRI/Bevacizumab (BEV) in Participants With Previously Treated Advanced Inoperable Metastatic Colorectal Cancer (mCRC)
Acronym: ELEVATE CRC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-587-6156; 2022-500177-13 (Other: European Medicines Agency)
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — magrolimab; Bevacizumab; Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI (Experimental): Participants will receive magrolimab + bevacizumab + FOLFIRI as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, every week (QW) beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, every 2 weeks (Q2W) beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours, Q2W (Days 1 and 15) of every 28-day cycle.
  Interventions: Drug: Magrolimab; Drug: Bevacizumab; Drug: Irinotecan; Drug: Fluorouracil; Drug: Leucovorin
- Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI (Experimental): Participants will receive magrolimab + bevacizumab + FOLFIRI as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, QW beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, Q2W beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours, Q2W (Days 1 and 15) of every 28-day cycle.
  Interventions: Drug: Magrolimab; Drug: Bevacizumab; Drug: Irinotecan; Drug: Fluorouracil; Drug: Leucovorin
- Randomized Cohort: Bevacizumab + FOLFIRI (Active Comparator): Participants will receive bevacizumab + FOLFIRI as mentioned below:
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours, Q2W (Days 1 and 15) of every 28-day cycle.
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Magrolimab — Administered intravenous infusion
  Other Names: GS-4721
  Arms: Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI; Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI
Drug: Bevacizumab — Administered intravenous infusion
Drug: Irinotecan — Administered intravenous infusion
  Other Names: CAMPTOSAR®
Drug: Fluorouracil — Administered intravenous infusion
Drug: Leucovorin — Administered intravenous infusion

SUMMARY:
The goals of this clinical study are to learn more about the safety, tolerability and effectiveness of magrolimab in combination with bevacizumab and 5-fluorouracil, irinotecan, and leucovorin (FOLFIRI) in previously treated participants with advanced inoperable metastatic colorectal cancer (mCRC).

The primary objectives of this study are: (safety run-in cohort) to evaluate safety and tolerability, and the recommended Phase 2 dose (RP2D) and (randomized cohort) to evaluate the efficacy of magrolimab in combination with bevacizumab and 5-fluorouracil, irinotecan, and leucovorin (FOLFIRI) in previously treated participants with advanced inoperable metastatic colorectal cancer (mCRC).

ELIGIBILITY:
Key Inclusion Criteria:

* Previously treated individuals with inoperable metastatic colorectal cancer (mCRC) who are ineligible for checkpoint inhibitor therapy (microsatellite instability (MSI)-H or mismatch repair deficient (dMMR) and are excluded).
* Histologically or cytologically confirmed adenocarcinoma originating in the colon or rectum (excluding appendiceal and anal canal cancers) who have progressed on or after 1 prior systemic therapy in the setting where curative resection is not indicated. This therapy must have included chemotherapy based on 5-fluorouracil (5-FU) or capecitabine with oxaliplatin and either bevacizumab, or for individuals with rat sarcoma (RAS) wild-type and left-sided tumors, bevacizumab, cetuximab, or panitumumab.
* Measurable disease (Response Evaluation Criteria in Solid Tumors (RECIST) V1.1 criteria).
* Individuals must have an eastern cooperative oncology group (ECOG) performance status of 0 or 1.
* Life expectancy of at least 12 weeks.
* Laboratory measurements, blood counts: adequate hemoglobin, neutrophil, and platelet counts
* Adequate liver function.
* Adequate renal function.

Key Exclusion Criteria:

* Prior anticancer therapy including chemotherapy, hormonal therapy, or investigational agents within 3 weeks or within at least 4 half-lives prior to magrolimab dosing (up to a maximum of 4 weeks), whichever is shorter.
* Known v-raf murine sarcoma viral oncogene homolog B1 gene mutation (BRAF V600E) or MSI-H mutations or dMMR.
* Persistent Grade 2 or more gastrointestinal bleeding.
* Individuals with prior irinotecan therapy.
* Clinically significant coronary artery disease or myocardial infarction within 6 months prior to inclusion.
* Peripheral neuropathy of more than Grade 2 (Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0).
* Known dihydropyrimidine dehydrogenase deficiency.
* Acute intestinal obstruction or sub-obstruction, history of inflammatory intestinal disease or extended resection of the small intestine. Presence of a colonic prosthesis.
* Unhealed wound, active gastric or duodenal ulcer, or bone fracture.
* History of abdominal fistulas, trachea-oesophageal fistulas, any other Grade 4 gastrointestinal perforations, nongastrointestinal fistulas, or intra-abdominal abscesses 6 months prior to screening.
* Uncontrolled arterial hypertension.
* Thromboembolic event in the 6 months before inclusion (eg, transitory ischemic stroke, stroke, subarachnoid hemorrhage) except peripheral deep vein thrombosis treated with anticoagulants.
* Active central nervous system (CNS) disease. Individuals with asymptomatic and stable, treated CNS lesions (radiation and/or surgery and/or other CNS-directed therapy who have not received corticosteroids for at least 4 weeks) are allowed.
* Red blood cell (RBC) transfusion dependence, defined as requiring more than 2 units of packed RBC transfusions during the 4-week period prior to screening.
* History of hemolytic anemia, autoimmune thrombocytopenia, or Evans syndrome in the last 3 months.
* Known hypersensitivity to any of the study drugs, the metabolites, or formulation excipient.
* Known inherited or acquired bleeding disorders.
* Significant disease or medical conditions, as assessed by the investigator and sponsor, that would substantially increase the risk-benefit ratio of participating in the study.
* Second malignancy, except treated basal cell or localized squamous skin carcinomas, or localized prostate cancer.
* Uncontrolled pleural effusion.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (51):
- United States (20):
  - City of Hope ( City of Hope National Medical Center, City of Hope Medical Center ), Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Torrance Memorial Physician Network, Redondo Beach, California
  - University of California Los Angeles (UCLA), Santa Monica, California
  - Orlando Health Cancer Institute, Orlando, Florida
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - University of Kansas, Westwood, Kansas
  - University of Michigan, Ann Arbor, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York, PC, East Syracuse, New York
  - AdventHealth, Rochester, New York
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Seattle Cancer Care Alliance (SCCA), Seattle, Washington
- Australia (8):
  - Westmead Hospital, Blacktown, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Southside Cancer Care Centre, Miranda, New South Wales
  - Genesis Care North Shore, St Leonards, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Belgium (2):
  - Hôpital de Jolimont, Haine-Saint-Paul
  - Centre Hospitalizer De L'Ardenne, Libramont-Chevigny
- Canada (2):
  - The Ottawa Hospital Cancer Centre, Ottawa
  - Princess Margaret Cancer Centre, Toronto
- France (4):
  - Centre Hospitalier Regional Universitaire Hopital Besancon, BesanÃ§on
  - Centre Léon Bérard - Centre de Lutte contre le Cancer, Lyon
  - Hopital franco brittanique, Paris
  - CHU de Tours, Tours
- Germany (2):
  - Carl Gustav Carus Management GMBH, Dresden
  - Klinikum rechts der Isar der TU Munchen Zentrum fur klinische Studien der Klinik und Poliklinik fur Innere Medizin III, München
- Hong Kong (2):
  - Hong Kong Integrated Oncology Centre, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Italy (5):
  - Istituto Romagnolo per lo Studio dei Tumori "Dino Amadori" - Medical Oncology Department, Meldola
  - Istituto Oncologico Veneto (IOV)- IRCCS, Padua
  - Azienda Ospedaliera Universitaria Pisana- UO Oncologia Medica, Pisa
  - Istituto di Ricovero e Cura a Carattere Scientifico - Istituto Clinico Humanitas, San Giovanni Rotondo
  - San Bortolo General Hospital- Oncology Department, Vicenza
- Pan American Center for Oncology Trials, LLC, San Juan, PR, Puerto Rico
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Català d'Oncologia- Hospital Duran I Reynals, L'Hospitalet de Llobregat
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital HM Sanchinarro, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fakih MG, Tejani M, Ren X, Landes D, Werneke S, Curtis KK et al. 439TiP A phase II (ph2), randomized study of magrolimab with bevacizumab and FOLFIRI in previously treated patients with advanced inoperable metastatic colorectal cancer (mCRC). Annals of Oncology 2022; 33(7):S735.
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-587-6156

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 124 participants were screened.
Pre-assignment Details: Participants were enrolled at study sites in Australia, Belgium, Canada, France, Germany, Hong Kong, Italy, Spain, the United States and Puerto Rico.
Groups:
- Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI: Participants received magrolimab + bevacizumab + FOLFIRI intravenous infusions for 36 weeks as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, every week (QW) beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, every 2 weeks (Q2W) beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m² IV bolus on first day, followed by 2400 mg/m² over the next 46 hours Q2W (Days 1 and 15) of every 28-day cycle.
- Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI: Participants received magrolimab + bevacizumab + FOLFIRI intravenous infusions for 34 weeks as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, QW beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, Q2W beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours, Q2W (Days 1 and 15) of every 28-day cycle.
- Randomized Cohort: Bevacizumab + FOLFIRI: Participants received bevacizumab + FOLFIRI intravenous infusions for 34 weeks as mentioned below:
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours Q2W (Days 1 and 15) of every 28-day cycle.
Period: Overall Study
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Started | 10 | 44 | 23
Completed | 0 | 0 | 0
Not Completed | 10 | 44 | 23
Not completed — Study Terminated by Sponsor | 4 | 33 | 12
Not completed — Death | 5 | 2 | 4
Not completed — Withdrew Consent | 0 | 5 | 4
Not completed — Investigator's Discretion | 0 | 1 | 3
Not completed — Subject Decision | 1 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening.
Groups:
- Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI: Participants received magrolimab + bevacizumab + FOLFIRI intravenous infusions for 36 weeks as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, every week (QW) beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, every 2 weeks (Q2W) beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours Q2W (Days 1 and 15) of every 28-day cycle.
- Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI: Participants received magrolimab + bevacizumab + FOLFIRI intravenous infusions for 34 weeks as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, QW beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, Q2W beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours Q2W (Days 1 and 15) of every 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI | Total
Number analyzed (Participants) | 10 | 44 | 23 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 31 | 18 | 58
  >=65 years | 1 | 13 | 5 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (11.1) | 59 (10.1) | 56 (13.1) | 57 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 17 | 9 | 32
  Male | 4 | 27 | 14 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 7 | 2 | 9
  Not Hispanic or Latino | 10 | 34 | 21 | 65
  Unknown or Not Reported | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 1 | 6
  White | 9 | 31 | 19 | 59
  More than one race | 0 | 2 | 1 | 3
  Unknown or Not Reported | 0 | 2 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 16 | 10 | 32
  Australia | 4 | 6 | 1 | 11
  Spain | 0 | 6 | 5 | 11
  Puerto Rico | 0 | 4 | 1 | 5
  Belgium | 0 | 3 | 2 | 5
  Italy | 0 | 2 | 3 | 5
  Canada | 0 | 3 | 0 | 3
  France | 0 | 3 | 0 | 3
  Germany | 0 | 1 | 0 | 1
  Hong Kong | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in Cohort: Number of Participants Experiencing Dose-limiting Toxicities (DLTs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: DLT was defined as any,
  * Grade 3 or higher hematologic toxicity including, serious hemolytic anemia, grade 4 neutropenia lasting > 7 days
  * An event meeting Hy's Law criteria:
    * Treatment-emergent alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation (≥ 3 x ULN) and,
    * Treatment-emergent total bilirubin elevation (> 2 x ULN), and absence of cholestasis (defined as alkaline phosphatase < 2 x ULN), and
    * No other good explanation for the injury (hepatitis A, B, C, or other viral hepatic injury, alcohol ingestion, congestive heart failure, worsening liver metastases, hemolysis))
  * Grade 3 or higher nonhematologic toxicity that has worsened in severity from pretreatment baseline during the DLT-assessment period
  * Grade 3 fatigue lasting > 7 days
  * In the opinion of the investigator, the AE was at least possibly related to magrolimab
Time Frame: First dose date up to 28 days
Population: Participants in DLT-Evaluable Analysis Set were analyzed. DLT-Evaluable Analysis Set was defined as all participants in Safety Run-in cohort who met one of the following criteria in the DLT-evaluable period (defined as the first 28 days):
  * Participant experienced a DLT at any time after initiation of first infusion of magrolimab.
  * Participant did not experience a DLT and completes at least 3 infusions of magrolimab and at least 2 doses of bevacizumab and FOLFIRI in Safety Run-in Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Safety Run-in Cohort: Percentage of Participants Experiencing Adverse Events (AEs) According to the NCI-CTCAE Version 5.0
Description: Treatment-emergent adverse events (TEAEs) were defined as any AE that begun on or after the date of first dose of study drug up to the date of last dose of study treatment plus 30 days or the day before initiation of subsequent anticancer therapy, whichever came first. An AE was any untoward medical occurrence in a clinical study participant administered a study drug that did not necessarily have a causal relationship with the treatment.
Time Frame: First dose date up to last dose date (up to 36 weeks) plus 30 days
Population: Participants in the Safety Run-in Cohort in the Safety Analysis Set were analyzed. The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Measure: Number; unit: percentage of participants
Groups:
- Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI: Participants received magrolimab + bevacizumab + FOLFIRI intravenous infusions for 36 weeks as mentioned below:
  * Magrolimab 1 mg/kg on Cycle 1 Day 1; 30 mg/kg, QW beginning at Day 8 and for the next 6 doses (Cycle 1 Days 8, 15, and 22, and Cycle 2 Days 1, 8, 15, and 22); 30 mg/kg, Q2W beginning 1 week after the last weekly 30 mg/kg dose (starting Cycle 3 Day 1 onwards) for every 28-day cycle.
  * Bevacizumab: 5 mg/kg, Q2W (Days 1 and 15) of every 28-day cycle.
  * FOLFIRI (Irinotecan 180 mg/m^2 + leucovorin 400 mg/m^2 + fluorouracil 400 mg/m^2 IV bolus on first day, followed by 2400 mg/m^2 over the next 46 hours Q2W (Days 1 and 15) of every 28-day cycle.
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI
Number analyzed (Participants) | 10
percentage of participants | 100.0

3. Primary Outcome: Safety Run-in Cohort: Percentage of Participants Experiencing Laboratory Abnormalities According to NCI-CTCAE Version 5.0
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least 1 toxicity grade after the date of first dose of study drug up to the date of last dose of study treatment plus 30 days or the day before initiation of subsequent anticancer therapy, whichever came first.
Time Frame: First dose date up to last dose date (up to 36 weeks) plus 30 days
Population: Participants in the Safety Run-in Cohort in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI
Number analyzed (Participants) | 10
percentage of participants
  Any Grade 1 or Higher | 100.0
  Grade 3 or 4 | 90.0

4. Primary Outcome: Randomized Cohort: Progression-free Survival (PFS) as Determined by Investigator Assessment Using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: PFS was defined as the time from the date of randomization until the earliest date of documented disease progression (PD) as determined by investigator assessment using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST V1.1), or death from any cause, whichever occurred first. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Kaplan-Meier (KM) estimates were used in outcome measure analysis.
Time Frame: Up to 83.4 weeks
Population: Participants in the Randomized Cohorts in the Intent-to-treat Analysis Set were analyzed. Intent-to-treat Analysis Set included all participants who were randomized in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 44 | 23
months | 6.2 [6.0 to NA] — Upper limit of confidence interval (CI) was not estimable due to low number of participants with events. | 6.7 [3.9 to NA] — Upper limit of CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI vs Randomized Cohort: Bevacizumab + FOLFIRI; Test type: Superiority; p = 0.9323, Unstratified Log-rank Test; 2-Sided P-value was based on unstratified log-rank test; Hazard Ratio (HR) = 0.956, 95% CI 2-sided [0.339 to 2.691] — Hazard ratio and its 95% CI were calculated using unstratified Cox proportional hazards regression model

5. Secondary Outcome: Randomized Cohort: Objective Response Rate (ORR) as Determined by Investigator Assessment Using RECIST Version 1.1
Description: ORR was defined as the percentage of participants who achieve complete response (CR) or partial response (PR) that was confirmed at least 4 weeks after initial documentation of response, as determined by investigator assessment per RECIST, Version 1.1. CR was defined as disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Clopper-Pearson estimates were used in outcome measure analysis. Percentages were rounded off.
Time Frame: Up to 83.4 weeks
Population: Participants in the Randomized Cohorts in the Intent-to-Treat Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 44 | 23
percentage of participants | 13.6 [5.2 to 27.4] | 0.0 [0.0 to 14.8]

6. Secondary Outcome: Randomized Cohort: Duration of Response (DOR) as Determined by Investigator Assessment Per RECIST Version 1.1
Description: DOR was defined as time from first documentation of CR or PR to the earliest date of documented disease progression as determined by investigator assessment, per RECIST V1.1, or death from any cause, whichever occurred first. PD was defined in outcome measure #4. CR and PR were defined in outcome measure #5.
  KM estimates were used in outcome measure analysis.
Time Frame: Up to 83.4 weeks
Population: Participants in the Randomized Cohorts in the Intent-to-Treat Analysis Set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 6 | 0
months | NA [NA to NA] — Median, lower and upper limit of CI were not estimable due to low number of participants with events. |

7. Secondary Outcome: Randomized Cohort: Overall Survival (OS)
Description: OS was defined as time from date of randomization to death from any cause. KM estimates were used in outcome measure analysis.
Time Frame: Up to 83.4 weeks
Population: Participants in the Randomized Cohort in the Intent-to-Treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 44 | 23
months | NA [NA to NA] — Median, lower and upper limit of CI were not estimable due to low number of participants with events. | 8.2 [6.1 to NA] — Upper limit of CI were not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI vs Randomized Cohort: Bevacizumab + FOLFIRI; Test type: Superiority; Hazard Ratio (HR) = 0.299, 95% CI 2-sided [0.056 to 1.600] — Hazard ratio and its 95% CI were calculated using unstratified Cox proportional hazards regression model

8. Secondary Outcome: Randomized Cohort: Change From Baseline of European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QLQ) - Core Questionnaire EORTC-QLQ-C30 Score
Description: EORTC QLQ-C30 is a quality of life (QOL) questionnaire for cancer participants, that has 30 items. 5 functional scales (physical, role, emotional, cognitive, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, loss of appetite, constipation, diarrhea, and financial difficulties). Scoring of the QLQ-C30 was performed according to QLQ-C30 Scoring manual. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the participant), while higher scores on the symptom and single-item scales indicated a higher level of symptoms (i.e. a worse state of the participant).
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4 and last cycle (Cycle 8) (Each cycle was of 28 days)
Population: Participants in the Randomized cohort in the Intent-to-treat Analysis Set with available data were analyzed. Data was collected until Cycle 8.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 38 | 18
Score on a scale
  Global Health Status / QoL: Baseline | 68.0 (20.1) | 69.0 (18.0)
  Global Health Status / QoL: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Global Health Status / QoL: Change from Baseline at Cycle 2 Day 1 | -1.3 (20.9) | -2.1 (17.1)
  Global Health Status / QoL: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Global Health Status / QoL: Change from Baseline at Cycle 3 Day 1 | 1.7 (17.8) | 5.4 (15.2)
  Global Health Status / QoL: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Global Health Status / QoL: Change from Baseline at Cycle 4 Day 1 | 0.4 (19.8) | -3.8 (13.6)
  Global Health Status / QoL: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Global Health Status / QoL: Change from Baseline at Cycle 8 Day 1 | 0.0 (23.6) | -16.7 (NA) — Standard deviation cannot be calculated for one participant.
  Functional Scales: Physical Functioning: Baseline | 83.5 (16.8) | 85.2 (15.3)
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 2 Day 1 | -5.7 (11.9) | -0.8 (6.4)
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 3 Day 1 | -0.8 (13.9) | -0.5 (4.9)
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Functional Scales: Physical Functioning: Change from Baseline at Cycle 4 Day 1 | -3.2 (8.1) | 0.0 (11.2)
  Functional Scales: Physical Functioning: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Functional Scales: Physical Functioning: Cycle 8 Day 1 | 0.0 (0.0) | -26.7 (NA) — Standard deviation cannot be calculated for one participant.
  Functional Scales: Role Functioning: Baseline | 74.1 (24.4) | 88.9 (15.1)
  Functional Scales: Role Functioning: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Functional Scales: Role Functioning: Change from Baseline at Cycle 2 Day 1 | -3.5 (19.9) | -13.5 (22.9)
  Functional Scales: Role Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Functional Scales: Role Functioning: Change from Baseline at Cycle 3 Day 1 | 3.3 (25.5) | -6.0 (16.8)
  Functional Scales: Role Functioning: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Functional Scales: Role Functioning: Change from Baseline at Cycle 4 Day 1 | -1.6 (16.6) | -10.6 (22.7)
  Functional Scales: Role Functioning: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Functional Scales: Role Functioning: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | -100.0 (NA) — Standard deviation cannot be calculated for one participant.
  Functional Scales: Emotional Functioning: Baseline | 75.4 (19.6) | 71.3 (23.4)
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 2 Day 1 | 9.1 (15.2) | 6.3 (17.3)
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 3 Day 1 | 8.0 (9.2) | 10.7 (14.8)
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 4 Day 1 | 5.6 (12.5) | 6.8 (18.2)
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Functional Scales: Emotional Functioning: Change from Baseline at Cycle 8 Day 1 | 12.5 (5.9) | 0.0 (NA) — Standard deviation cannot be calculated for one participant.
  Functional Scales: Cognitive Functioning: Baseline | 89.9 (15.3) | 88.0 (17.0)
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 2 Day 1 | -0.5 (12.1) | -2.1 (17.1)
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 3 Day 1 | 0.7 (17.7) | 2.4 (17.1)
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 4 Day 1 | -4.0 (19.7) | -3.0 (10.1)
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Functional Scales: Cognitive Functioning: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | 16.7 (NA) — Standard deviation cannot be calculated for one participant.
  Functional Scales: Social Functioning: Baseline | 71.5 (21.9) | 82.4 (25.2)
  Functional Scales: Social Functioning: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Functional Scales: Social Functioning: Change from Baseline at Cycle 2 Day 1 | 2.0 (24.2) | 1.0 (18.7)
  Functional Scales: Social Functioning: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Functional Scales: Social Functioning: Change from Baseline at Cycle 3 Day 1 | 6.0 (25.4) | -3.6 (16.2)
  Functional Scales: Social Functioning: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Functional Scales: Social Functioning: Change from Baseline at Cycle 4 Day 1 | 4.0 (16.6) | 1.5 (13.9)
  Functional Scales: Social Functioning: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Functional Scales: Social Functioning: Change from Baseline at Cycle 8 Day 1 | 8.3 (11.8) | -50.0 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Fatigue: Baseline | 31.0 (22.1) | 24.1 (16.3)
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 2 Day 1 | 7.7 (19.7) | 4.2 (16.2)
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 3 Day 1 | 4.9 (20.1) | 1.6 (17.4)
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 4 Day 1 | 5.8 (16.3) | 7.1 (15.1)
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Fatigue: Change from Baseline at Cycle 8 Day 1 | -5.6 (39.3) | 55.6 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Nausea and Vomiting: Baseline | 4.8 (11.6) | 3.7 (10.8)
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 2 Day 1 | 6.1 (18.1) | 11.5 (18.0)
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 3 Day 1 | 3.3 (8.3) | 3.6 (9.6)
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 4 Day 1 | 6.3 (11.2) | 3.0 (6.7)
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Nausea and Vomiting: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | 16.7 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Pain: Baseline | 23.7 (23.8) | 19.4 (29.8)
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 2 Day 1 | -4.0 (18.6) | 0.0 (17.2)
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 3 Day 1 | -6.7 (19.2) | -11.9 (20.1)
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 4 Day 1 | -1.6 (19.7) | -9.1 (17.3)
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Pain: Change from Baseline at Cycle 8 Day 1 | -16.7 (0.0) | 33.3 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Dyspnoea: Baseline | 7.9 (18.1) | 9.3 (15.4)
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 2 Day 1 | 11.1 (28.5) | 2.1 (14.8)
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 3 Day 1 | 5.3 (12.5) | -2.4 (8.9)
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 4 Day 1 | 11.1 (16.1) | 6.1 (13.5)
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Dyspnoea: Change from Baseline at Cycle 8 Day 1 | 16.7 (23.6) | 33.3 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Insomnia: Baseline | 29.8 (31.8) | 31.5 (29.1)
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 2 Day 1 | -4.0 (20.0) | -2.1 (19.1)
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 3 Day 1 | -5.3 (22.9) | -7.1 (29.8)
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 4 Day 1 | -3.2 (25.6) | -12.1 (30.8)
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Insomnia: Change from Baseline at Cycle 8 Day 1 | -16.7 (70.7) | 0.0 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Appetite Loss: Baseline | 21.1 (28.4) | 11.1 (22.9)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 2 Day 1 | 5.1 (20.6) | 6.2 (21.8)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 3 Day 1 | 5.3 (22.9) | 2.4 (20.5)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 4 Day 1 | 1.6 (24.7) | 9.1 (21.6)
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Appetite Loss: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | 33.3 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Constipation: Baseline | 7.9 (18.1) | 13.0 (25.9)
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 2 Day 1 | 12.1 (26.1) | 2.1 (25.7)
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 3 Day 1 | 14.7 (25.6) | 0.0 (37.0)
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 4 Day 1 | 12.7 (24.7) | 6.1 (25.0)
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Constipation: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | 66.7 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Diarrhoea: Baseline | 14.0 (24.1) | 5.6 (12.8)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 2 Day 1 | 12.1 (20.1) | 16.7 (21.1)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 3 Day 1 | 5.3 (26.7) | 16.7 (17.3)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 4 Day 1 | 9.5 (26.1) | 15.2 (17.4)
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Diarrhoea: Change from Baseline at Cycle 8 Day 1 | 33.3 (0.0) | 66.7 (NA) — Standard deviation cannot be calculated for one participant.
  Symptom Scales / Items: Financial Difficulties: Baseline | 26.3 (35.6) | 13.0 (23.3)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 33 | 16
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 2 Day 1 | -6.1 (24.2) | 2.1 (8.3)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 14
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 3 Day 1 | -8.0 (24.1) | 7.1 (19.3)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 11
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 4 Day 1 | -3.2 (25.6) | 3.0 (10.1)
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Symptom Scales / Items: Financial Difficulties: Change from Baseline at Cycle 8 Day 1 | 0.0 (0.0) | 0.0 (NA) — Standard deviation cannot be calculated for one participant.

9. Secondary Outcome: Randomized Cohort: Number of Participants With 5-level EuroQol 5 Dimensions Questionnaire (EQ-5D-5L) Score
Description: EQ-5D-5L was an instrument for use as a measure of health outcome. The EQ-5D-5L consisted of 2 sections: EuroQoL (5 dimensions) (EQ-5D) descriptive system and the EuroQoL visual analogue scale (EQ-VAS). EQ-5D comprised the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension had 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Number of participants per category were reported.
Time Frame: Day 1 of Cycles 2, 3, 4 and last cycle (Cycle 8) (Each cycle is of 28 days)
Population: Participants in the Randomized Cohort in the Intent-to-treat Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 38 | 17
Participants
  Mobility: Baseline: No Problems | 27 | 12
  Mobility: Baseline: Slight Problems | 5 | 4
  Mobility: Baseline: Moderate Problems | 5 | 1
  Mobility: Baseline: Severe Problems | 1 | 0
  Mobility: Baseline: Extreme Problems | 0 | 0
  Mobility: Cycle 2 Day 1: number analyzed (Participants) | 31 | 17
  Mobility: Cycle 2 Day 1: No Problems | 21 | 10
  Mobility: Cycle 2 Day 1: Slight Problems | 6 | 6
  Mobility: Cycle 2 Day 1: Moderate Problems | 4 | 1
  Mobility: Cycle 2 Day 1: Severe Problems | 0 | 0
  Mobility: Cycle 2 Day 1: Extreme Problems | 0 | 0
  Mobility: Cycle 3 Day 1: number analyzed (Participants) | 25 | 16
  Mobility: Cycle 3 Day 1: No Problems | 20 | 9
  Mobility: Cycle 3 Day 1: Slight Problems | 3 | 7
  Mobility: Cycle 3 Day 1: Moderate Problems | 2 | 0
  Mobility: Cycle 3 Day 1: Severe Problems | 0 | 0
  Mobility: Cycle 3 Day 1: Extreme Problems | 0 | 0
  Mobility: Cycle 4 Day 1: number analyzed (Participants) | 22 | 12
  Mobility: Cycle 4 Day 1: No Problems | 15 | 10
  Mobility: Cycle 4 Day 1: Slight Problems | 3 | 2
  Mobility: Cycle 4 Day 1: Moderate Problems | 4 | 0
  Mobility: Cycle 4 Day 1: Severe Problems | 0 | 0
  Mobility: Cycle 4 Day 1: Extreme Problems | 0 | 0
  Mobility: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Mobility: Cycle 8 Day 1: No Problems | 2 | 0
  Mobility: Cycle 8 Day 1: Slight Problems | 0 | 1
  Mobility: Cycle 8 Day 1: Moderate Problems | 0 | 0
  Mobility: Cycle 8 Day 1: Severe Problems | 0 | 0
  Mobility: Cycle 8 Day 1: Extreme Problems | 0 | 0
  Self-Care: Baseline: No Problems | 32 | 17
  Self-Care: Baseline: Slight Problems | 4 | 0
  Self-Care: Baseline: Moderate Problems | 1 | 0
  Self-Care: Baseline: Severe Problems | 0 | 0
  Self-Care: Baseline: Extreme Problems | 1 | 0
  Self-Care: Cycle 2 Day 1: number analyzed (Participants) | 31 | 17
  Self-Care: Cycle 2 Day 1: No Problems | 25 | 15
  Self-Care: Cycle 2 Day 1: Slight Problems | 5 | 2
  Self-Care: Cycle 2 Day 1: Moderate Problems | 1 | 0
  Self-Care: Cycle 2 Day 1: Severe Problems | 0 | 0
  Self-Care: Cycle 2 Day 1: Extreme Problems | 0 | 0
  Self-Care: Cycle 3 Day 1: number analyzed (Participants) | 25 | 16
  Self-Care: Cycle 3 Day 1: No Problems | 24 | 16
  Self-Care: Cycle 3 Day 1: Slight Problems | 0 | 0
  Self-Care: Cycle 3 Day 1: Moderate Problems | 0 | 0
  Self-Care: Cycle 3 Day 1: Severe Problems | 0 | 0
  Self-Care: Cycle 3 Day 1: Extreme Problems | 1 | 0
  Self-Care: Cycle 4 Day 1: number analyzed (Participants) | 22 | 12
  Self-Care: Cycle 4 Day 1: No Problems | 20 | 11
  Self-Care: Cycle 4 Day 1: Slight Problems | 0 | 1
  Self-Care: Cycle 4 Day 1: Moderate Problems | 2 | 0
  Self-Care: Cycle 4 Day 1: Severe Problems | 0 | 0
  Self-Care: Cycle 4 Day 1: Extreme Problems | 0 | 0
  Self-Care: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Self-Care: Cycle 8 Day 1: No Problems | 2 | 1
  Self-Care: Cycle 8 Day 1: Slight Problems | 0 | 0
  Self-Care: Cycle 8 Day 1: Moderate Problems | 0 | 0
  Self-Care: Cycle 8 Day 1: Severe Problems | 0 | 0
  Self-Care: Cycle 8 Day 1: Extreme Problems | 0 | 0
  Usual Activities: Baseline: No Problems | 18 | 11
  Usual Activities: Baseline: Slight Problems | 14 | 3
  Usual Activities: Baseline: Moderate Problems | 6 | 2
  Usual Activities: Baseline: Severe Problems | 0 | 0
  Usual Activities: Baseline: Extreme Problems | 0 | 1
  Usual Activities: Cycle 2 Day 1: number analyzed (Participants) | 31 | 17
  Usual Activities: Cycle 2 Day 1: No Problems | 15 | 10
  Usual Activities: Cycle 2 Day 1: Slight Problems | 11 | 5
  Usual Activities: Cycle 2 Day 1: Moderate Problems | 4 | 2
  Usual Activities: Cycle 2 Day 1: Severe Problems | 1 | 0
  Usual Activities: Cycle 2 Day 1: Extreme Problems | 0 | 0
  Usual Activities: Cycle 3 Day 1: number analyzed (Participants) | 25 | 16
  Usual Activities: Cycle 3 Day 1: No Problems | 17 | 9
  Usual Activities: Cycle 3 Day 1: Slight Problems | 7 | 5
  Usual Activities: Cycle 3 Day 1: Moderate Problems | 1 | 1
  Usual Activities: Cycle 3 Day 1: Severe Problems | 0 | 1
  Usual Activities: Cycle 3 Day 1: Extreme Problems | 0 | 0
  Usual Activities: Cycle 4 Day 1: number analyzed (Participants) | 22 | 12
  Usual Activities: Cycle 4 Day 1: No Problems | 13 | 10
  Usual Activities: Cycle 4 Day 1: Slight Problems | 6 | 2
  Usual Activities: Cycle 4 Day 1: Moderate Problems | 3 | 0
  Usual Activities: Cycle 4 Day 1: Severe Problems | 0 | 0
  Usual Activities: Cycle 4 Day 1: Extreme Problems | 0 | 0
  Usual Activities: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Usual Activities: Cycle 8 Day 1: No Problems | 2 | 1
  Usual Activities: Cycle 8 Day 1: Slight Problems | 0 | 0
  Usual Activities: Cycle 8 Day 1: Moderate Problems | 0 | 0
  Usual Activities: Cycle 8 Day 1: Severe Problems | 0 | 0
  Usual Activities: Cycle 8 Day 1: Extreme Problems | 0 | 0
  Pain/Discomfort: Baseline: No Problems | 14 | 10
  Pain/Discomfort: Baseline: Slight Problems | 15 | 2
  Pain/Discomfort: Baseline: Moderate Problems | 7 | 4
  Pain/Discomfort: Baseline: Severe Problems | 2 | 1
  Pain/Discomfort: Baseline: Extreme Problems | 0 | 0
  Pain/Discomfort: Cycle 2 Day 1: number analyzed (Participants) | 31 | 17
  Pain/Discomfort: Cycle 2 Day 1: No Problems | 16 | 9
  Pain/Discomfort: Cycle 2 Day 1: Slight Problems | 9 | 3
  Pain/Discomfort: Cycle 2 Day 1: Moderate Problems | 5 | 4
  Pain/Discomfort: Cycle 2 Day 1: Severe Problems | 1 | 1
  Pain/Discomfort: Cycle 2 Day 1: Extreme Problems | 0 | 0
  Pain/Discomfort: Cycle 3 Day 1: number analyzed (Participants) | 25 | 16
  Pain/Discomfort: Cycle 3 Day 1: No Problems | 14 | 10
  Pain/Discomfort: Cycle 3 Day 1: Slight Problems | 11 | 3
  Pain/Discomfort: Cycle 3 Day 1: Moderate Problems | 0 | 3
  Pain/Discomfort: Cycle 3 Day 1: Severe Problems | 0 | 0
  Pain/Discomfort: Cycle 3 Day 1: Extreme Problems | 0 | 0
  Pain/Discomfort: Cycle 4 Day 1: number analyzed (Participants) | 22 | 12
  Pain/Discomfort: Cycle 4 Day 1: No Problems | 13 | 8
  Pain/Discomfort: Cycle 4 Day 1: Slight Problems | 6 | 4
  Pain/Discomfort: Cycle 4 Day 1: Moderate Problems | 2 | 0
  Pain/Discomfort: Cycle 4 Day 1: Severe Problems | 1 | 0
  Pain/Discomfort: Cycle 4 Day 1: Extreme Problems | 0 | 0
  Pain/Discomfort: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Pain/Discomfort: Cycle 8 Day 1: No Problems | 2 | 0
  Pain/Discomfort: Cycle 8 Day 1: Slight Problems | 0 | 0
  Pain/Discomfort: Cycle 8 Day 1: Moderate Problems | 0 | 1
  Pain/Discomfort: Cycle 8 Day 1: Severe Problems | 0 | 0
  Pain/Discomfort: Cycle 8 Day 1: Extreme Problems | 0 | 0
  Anxiety/Depression: Baseline: No Problems | 25 | 7
  Anxiety/Depression: Baseline: Slight Problems | 10 | 9
  Anxiety/Depression: Baseline: Moderate Problems | 2 | 1
  Anxiety/Depression: Baseline: Severe Problems | 1 | 0
  Anxiety/Depression: Baseline: Extreme Problems | 0 | 0
  Anxiety/Depression: Cycle 2 Day 1: number analyzed (Participants) | 31 | 17
  Anxiety/Depression: Cycle 2 Day 1: No Problems | 21 | 9
  Anxiety/Depression: Cycle 2 Day 1: Slight Problems | 9 | 4
  Anxiety/Depression: Cycle 2 Day 1: Moderate Problems | 1 | 4
  Anxiety/Depression: Cycle 2 Day 1: Severe Problems | 0 | 0
  Anxiety/Depression: Cycle 2 Day 1: Extreme Problems | 0 | 0
  Anxiety/Depression: Cycle 3 Day 1: number analyzed (Participants) | 25 | 16
  Anxiety/Depression: Cycle 3 Day 1: No Problems | 15 | 12
  Anxiety/Depression: Cycle 3 Day 1: Slight Problems | 8 | 2
  Anxiety/Depression: Cycle 3 Day 1: Moderate Problems | 2 | 1
  Anxiety/Depression: Cycle 3 Day 1: Severe Problems | 0 | 1
  Anxiety/Depression: Cycle 3 Day 1: Extreme Problems | 0 | 0
  Anxiety/Depression: Cycle 4 Day 1: number analyzed (Participants) | 22 | 12
  Anxiety/Depression: Cycle 4 Day 1: No Problems | 11 | 7
  Anxiety/Depression: Cycle 4 Day 1: Slight Problems | 11 | 4
  Anxiety/Depression: Cycle 4 Day 1: Moderate Problems | 0 | 1
  Anxiety/Depression: Cycle 4 Day 1: Severe Problems | 0 | 0
  Anxiety/Depression: Cycle 4 Day 1: Extreme Problems | 0 | 0
  Anxiety/Depression: Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Anxiety/Depression: Cycle 8 Day 1: No Problems | 2 | 0
  Anxiety/Depression: Cycle 8 Day 1: Slight Problems | 0 | 0
  Anxiety/Depression: Cycle 8 Day 1: Moderate Problems | 0 | 1
  Anxiety/Depression: Cycle 8 Day 1: Severe Problems | 0 | 0
  Anxiety/Depression: Cycle 8 Day 1: Extreme Problems | 0 | 0

10. Secondary Outcome: Randomized Cohort: Change From Baseline in the EuroQoL Visual Analogue Scale (EQ-VAS) Score
Description: The EQ-VAS recorded the participants' self-rated health on a vertical VAS, where the end points were labeled "the best health you can imagine" and "the worst health you can imagine." The scale range from 0 to 100, where '100' rating denotes the best health and '0' rating denotes the worst health. The EQ-VAS is used as a quantitative measure of health outcome that reflects the participants' own judgment.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4 and last cycle (Cycle 8) (Each cycle is of 28 days)
Population: Participants in the Randomized Cohort in the Intent-to-treat Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 38 | 17
Units on a scale
  Baseline | 72.2 (17.58) | 75.9 (12.78)
  Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 30 | 15
  Change from Baseline at Cycle 2 Day 1 | -3.0 (14.97) | -4.8 (17.55)
  Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 13
  Change from Baseline at Cycle 3 Day 1 | 3.6 (17.47) | -4.5 (15.14)
  Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 9
  Change from Baseline at Cycle 4 Day 1 | -0.3 (16.63) | -3.7 (12.32)
  Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 1
  Change from Baseline at Cycle 8 Day 1 | 5.0 (7.07) | -44.0 (NA) — Standard deviation cannot be calculated for one participant.

11. Secondary Outcome: Randomized Cohort: Change From Baseline of the Functional Assessment of Cancer Therapy (FACT) Colorectal Symptom Index (FCSI) Score
Description: The FCSI was a set of brief, clinically relevant, colorectal cancer symptoms for assessing symptomatic response. It comprised the most important symptoms associated with colorectal cancer, including energy, pain, weight, diarrhea, nausea, swelling or cramps in the stomach area, appetite, ability to enjoy life, and overall quality of life. The 9 questions were combined in three algorithms to provide information for 3 domains: colorectal cancer symptoms, physical well-being, and functional well-being. Each of the 9 items were scored from "0" to "4" representing "Not at All" through to "Very Much True". The raw score for all items was transformed to a 0-100 scale, and the average for each of the 3 subscales was calculated; high scores illustrated an improved state.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4 and last cycle (Cycle 8) (Each cycle is of 28 days)
Population: Participants in the Randomized Cohort in the Intent-to-Treat Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
Number analyzed (Participants) | 38 | 17
Score on a scale
  FCSI Score: Baseline | 27.1 (5.8) | 27.8 (4.8)
  FCSI Score: Change from Baseline at Cycle 2 Day 1: number analyzed (Participants) | 30 | 15
  FCSI Score: Change from Baseline at Cycle 2 Day 1 | -1.1 (3.7) | -0.3 (3.4)
  FCSI Score: Change from Baseline at Cycle 3 Day 1: number analyzed (Participants) | 25 | 13
  FCSI Score: Change from Baseline at Cycle 3 Day 1 | -0.6 (3.5) | -0.9 (5.0)
  FCSI Score: Change from Baseline at Cycle 4 Day 1: number analyzed (Participants) | 21 | 9
  FCSI Score: Change from Baseline at Cycle 4 Day 1 | -0.6 (4.1) | 0.4 (4.6)
  FCSI Score: Change from Baseline at Cycle 8 Day 1: number analyzed (Participants) | 2 | 0
  FCSI Score: Change from Baseline at Cycle 8 Day 1 | -1.0 (2.8) |

12. Secondary Outcome: Safety Run-in and Randomized Cohorts: Magrolimab Concentration Versus Time
Time Frame: Predose: Day 15, 29, 57, 113 and 169; Postdose: Day 57 (1 hour)
Population: Participants in the Pharmacokinetic (PK) Analysis Set with available data were analyzed. The PK Analysis Set was defined as all participants who received any amount of magrolimab and have at least 1 measurable posttreatment serum concentration of magrolimab.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI
Number analyzed (Participants) | 9 | 36
μg/mL
  Day 15: Predose: number analyzed (Participants) | 2 | 35
  Day 15: Predose | 187 (41.7) | 186 (55.0)
  Day 29: Predose | 581 (270.0) | 412 (163.0)
  Day 57: Predose: number analyzed (Participants) | 7 | 24
  Day 57: Predose | 889 (236.0) | 610 (204.0)
  Day 57: 1 hour Postdose: number analyzed (Participants) | 6 | 25
  Day 57: 1 hour Postdose | 1850 (385.0) | 1220 (360.0)
  Day 113: Predose: number analyzed (Participants) | 6 | 18
  Day 113: Predose | 469 (134.0) | 310 (166.0)
  Day 169: Predose: number analyzed (Participants) | 3 | 8
  Day 169: Predose | 480 (95.8) | 295 (128.0)

13. Secondary Outcome: Safety Run-in and Randomized Cohorts: Percentage of Participants With Antidrug Antibodies (ADA) to Magrolimab
Time Frame: Up to 36 weeks
Population: Participants in the Immunogenicity Analysis Set with available data were analyzed. Immunogenicity Analysis Set included all participants who received any amount of magrolimab and had at least 1 evaluable anti-drug antibody test result.
Measure: Number; unit: percentage of participants
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI
Number analyzed (Participants) | 10 | 37
percentage of participants | 0.0 | 5.4

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to 83.4 weeks; Adverse events: Up to 36 weeks plus 30 days
Description: All-cause mortality: All Enrolled Analysis Set included all participants who received a study subject identification number in the study after screening. Adverse events: The Safety Analysis Set included all participants who took at least 1 dose of any study drug.
Arm/Group | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI | Randomized Cohort: Bevacizumab + FOLFIRI
All-Cause Mortality (participants affected / at risk) | 6/10 | 2/44 | 5/23
Serious Adverse Events (participants affected / at risk) | 5/10 | 16/44 | 6/21
Other Adverse Events (participants affected / at risk) | 10/10 | 43/44 | 19/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI (N=10) | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI (N=44) | Randomized Cohort: Bevacizumab + FOLFIRI (N=21)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Malignant gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 2 | 0 | 0
Rectourethral fistula (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Anal abscess (Infections and infestations) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vascular device infection (Infections and infestations) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Run-in Cohort: Magrolimab + Bevacizumab + FOLFIRI (N=10) | Randomized Cohort: Magrolimab + Bevacizumab + FOLFIRI (N=44) | Randomized Cohort: Bevacizumab + FOLFIRI (N=21)
Anaemia (Blood and lymphatic system disorders) | 6 | 25 | 4
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 13 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 0
Dry eye (Eye disorders) | 2 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 0
Vitreous floaters (Eye disorders) | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 3 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 10 | 4
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 9 | 5
Diarrhoea (Gastrointestinal disorders) | 6 | 25 | 11
Dry mouth (Gastrointestinal disorders) | 0 | 3 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 23 | 10
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal tenesmus (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 16 | 2
Vomiting (Gastrointestinal disorders) | 4 | 14 | 5
Asthenia (General disorders) | 0 | 9 | 3
Chest pain (General disorders) | 1 | 1 | 0
Chills (General disorders) | 1 | 6 | 1
Fatigue (General disorders) | 8 | 19 | 6
Influenza like illness (General disorders) | 1 | 1 | 2
Malaise (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 3 | 2
Pyrexia (General disorders) | 2 | 7 | 4
Subcapsular hepatic haematoma (Hepatobiliary disorders) | 1 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 2 | 1
Gingivitis (Infections and infestations) | 2 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 4 | 4 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 2
Stoma complication (Injury, poisoning and procedural complications) | 1 | 0 | 1
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 2 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 2 | 1
Lymphocyte count decreased (Investigations) | 1 | 6 | 1
Neutrophil count decreased (Investigations) | 4 | 10 | 5
Platelet count decreased (Investigations) | 3 | 7 | 1
Weight decreased (Investigations) | 1 | 6 | 4
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 9 | 2
Decreased appetite (Metabolism and nutrition disorders) | 4 | 15 | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 6 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 5 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 0 | 6 | 1
Dysgeusia (Nervous system disorders) | 1 | 4 | 2
Headache (Nervous system disorders) | 4 | 15 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 6 | 2
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 3 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 7 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 5
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 9 | 7
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 4 | 3
Hypotension (Vascular disorders) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2023-10-31): https://cdn.clinicaltrials.gov/large-docs/29/NCT05330429/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/29/NCT05330429/SAP_001.pdf